CLINICAL TRIAL: NCT05541536
Title: Facilitating Learning Health Care (LHC) and Neonatal Research: Effects of a Brief Introductory Discussion Between a Neonatologist and the Parents of Eligible Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Susan Wootton, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: QI Project No. 2022-1349
Record Dates: First submitted 2022-08-31; First posted 2022-09-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Understanding of Consent in Clinical Research; Implementation of Consent in Clinical Research

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General information pamphlet plus Consultation meeting (Experimental): Study team member will approach mothers < 24 hrs (up to 5 min prior) of CRC approach for NRN trial. During the consultation meeting (5 minutes), the study team member will review the pamphlet and answer any questions. Visits will ideally occur in person. If the mother is not at bedside, 1 attempt will be made to reach the mother by phone in which case the pamphlet will be forwarded by mail.
  Interventions: Other: Consultation meeting; Other: Pamphlet
- Usual Care (Active Comparator): Study participants will not receive the general information pamphlet or consultation.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Consultation meeting — Study team member will approach mothers < 24 hrs (up to 5 min prior) of CRC approach for NRN trial. During the consultation meeting (5 minutes), the study team member will review the pamphlet and answer any questions. Visits will ideally occur in person. If the mother is not at bedside, 1 attempt will be made to reach the mother by phone in which case the pamphlet will be forwarded by mail.
  Arms: General information pamphlet plus Consultation meeting
Other: Pamphlet — Study team member will distribute pamphlet to beside nurse to give to mother. The pamphlet provides information about Learning Health Care (LHC) and clinical research.
  Arms: General information pamphlet plus Consultation meeting
Other: Usual Care — Study participants will not receive the general information pamphlet or consultation.
  Arms: Usual Care

SUMMARY:
The primary purpose of this pilot quality improvement study is to assess the impact of a brief introductory discussion about Learning Health Care (LHC) and clinical research between a neonatologist and the mothers (and the fathers, if present) of infants eligible for trials of the Neonatal Research Network (NRN) before they are approached for consent by clinical research coordinator (CRC) approach for NRN trial). Mothers will also be given a general information pamphlet addressing the same topic.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants eligible for Neonatal Research Network (NRN) trial (antenatal or postnatal)
* English or Spanish speaking
* Available for in-person (preference) or phone consultation meeting
* Mother not already approached for NRN trial

Exclusion Criteria:

* Mother already approached by clinical research coordinator (CRC) for NRN trial

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Neonatal Research Network (NRN) trial consent rate | Within 1 week of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wootton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- McGovern Medical School at UTHealth Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No